CLINICAL TRIAL: NCT05955170
Title: Tucatinib in Combination With Oral Etoposide (VP16) - Trastuzumab in Patients With Metastatic HER2+ Breast Cancer After Progression Under Tucatinib-Capecitabine-Trastuzumab or Toxicity Related to Capecitabine: a Multicenter Phase II
Brief Title: Tucatinib in Combination With Oral Etoposide andTrastuzumab in Patients With Metastatic HER2+ Breast Cancer
Acronym: TUC-TOC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2021-06
Record Dates: First submitted 2023-07-04; First posted 2023-07-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — tucatinib; Trastuzumab

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, phase II study to evaluate the efficacy, safety, tolerability, pharmacokinetics of the combination of tucatinib-Oral VP16-trastuzumab in patients with HER2-positive metastatic breast cancer (HER2+ MBC) after progression on tucatinib-capecitabine-trastuzumab or capecitabine-related toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of tucatinib-Oral VP16-trastuzumab (Experimental): The safety run in part will be a safety evaluation including 6 patients at dose D of Oral VP16 per day, trastuzumab 600mg SC flat dose or 6mg/kg IV every 3 weeks and tucatinib 300mg PO BID.
  The evaluable population for DLT in this Part 1 is defined as patients who have completed the first 2 cycles of treatment (i.e.6 weeks) and received 100% of the planned dose of tucatinib-Oral VP16-trastuzumab.Patients treated at Dose Recommended during the safety run-in part will be considered as evaluable for the part II.
  Interventions: Drug: Tucatinib in Combination of Oral VP16 and trastuzumab

INTERVENTIONS:
Drug: Tucatinib in Combination of Oral VP16 and trastuzumab — Combination of tucatinib-Oral VP16-trastuzumab

SUMMARY:
This is an open-label, multicenter, phase II study to evaluate the efficacy, safety, tolerability, pharmacokinetics of the combination of tucatinib-Oral VP16-trastuzumab in patients with HER2-positive metastatic breast cancer (HER2+ MBC) after progression on tucatinib-capecitabine-trastuzumab or capecitabine-related toxicity.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II study to evaluate the efficacy, safety, tolerability, pharmacokinetics of the combination of tucatinib-Oral VP16-trastuzumab in patients with HER2-positive metastatic breast cancer (HER2+ MBC) after progression on tucatinib-capecitabine-trastuzumab or capecitabine-related toxicity.

The study has two sequential parts:

* Part 1 is a safety run-in part evaluating the safety of the combination to confirm the recommended dose;
* Part 2 will evaluate the efficacy of the combination at the recommended dose. Both parts will include patients with HER2 positive metastatic breast cancer.

In part 1, a D-dose is evaluated; only in case of unacceptable toxicity at the D-dose, a D-1 dose will be investigated.

In part 2, patients will be treated with oral VP16 at the dose recommended in part 1.

Dose reductions will be allowed on subsequent cycles in case of toxicity.

All enrolled patients will receive the combination of tucatinib, oral VP16, trastuzumab until disease progression, unacceptable toxicity, and withdrawal of patient consent, investigator decision, and loss to follow-up, death, patient non-compliance, or discontinuation of the study by the sponsor.

Tumor assessments should be performed according to RECIST v1.1 criteria at baseline and every 6 weeks (± 7 days) for the first 24 weeks, then every 9 weeks (± 7 days) until documented disease progression, withdrawal of consent, or death.

ELIGIBILITY:
Inclusion Criteria:

1. First disease progression under tucatinib-capecitabine-trastuzumab. OR Medical contra-indication to initiate or continue capecitabine in association with tucatinib-trastuzumab (investigator's decision based on patient medical history, DPD deficiency and/or capecitabine grade 2 toxicity or higher).
2. Age > 18 years,
3. Histologically confirmed HER2+ breast carcinoma (ASCO/CAP guidelines) with archived tumor tissue available,
4. Have a life expectancy of at least 3 months,
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1,
6. Participants must be able to swallow capsules,
7. Participants must be able and willing to be available for the duration of the study and are willing to follow study procedures,
8. Measurable disease, assessed by RECIST version 1,
9. Patients with brain metastases are eligible:

   * Unless urgent treatment is required
   * If time since WBRT is ≥ 21 days prior to first dose of treatment, time since SRS is ≥ 7 days prior to first dose of treatment, or time since surgical resection is ≥ 28 days
10. Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions
11. Left ventricular ejection fraction (LVEF) ≥ 50% (within 4 weeks before inclusion)
12. Adequate organ function (obtained within 14 days prior to treatment start) as evidenced by:

    o Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L

    o Hemoglobin (Hgb) ≥ 9 g/dL

    o Platelet count ≥ 100 X 10^9/L
    * Bilirubin ≤ 1.5 X upper limit of normal (ULN), except for patients with a documented history of Gilbert's disease (≤ 2 X ULN)
    * Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5 X ULN (for patients with liver metastases ≤ 5 X ULN);
    * Alkaline phosphatase (AP) ≤ 3 X ULN (for patients with liver metastases, ≤ 5 X ULN);
    * Serum creatinine ≤ 1.5 mg/dL (133 μmol/L) or calculated creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula).
13. If the patient is female:

Women of childbearing potential (WCBP): negative serum pregnancy test. The patient must be willing to use effective methods of contraception. Patients must be postmenopausal, surgically infertile, or willing to use a physical barrier method of contraception in addition to an intrauterine device or hormonal contraception until at least 6 months after completion of study treatment,

If the patient is male:

Male patients must agree to use an acceptable method of contraception (e.g., condom) during the study and for 3 months after completion of investigational treatment, 14. Patients must be covered by a health insurance plan. 15. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Have previously been treated with:

   a. lapatinib within 12 months of starting study treatment (except in cases where lapatinib was given for ≤ 21 days and was discontinued for reasons other than disease progression or severe toxicity) b. neratinib, afatinib, or other investigational HER2/ EGFR or HER2 TKI at any time previously (excepted for patients already under tucatinib who continue without interruption).
2. Patients who are pre-treated with tucatinib and who received a decreased dose of tucatinib (<300mg twice daily) are not eligible in the safety run-in phase.
3. Have used a strong CYP3A4 or CYP2C8 inhibitor within 5 half-lives of the inhibitor, or have used a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment (see Appendix 4 and 5)
4. Patients unable for any reason to undergo MRI of the brain.
5. Leptomeningeal metastases or brain metastases requiring immediate symptomatic treatment or a high dose of corticosteroid therapy (≥2mg/day dexamethasone or equivalent).
6. Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy
7. Any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1 at time of treatment start, with the following exceptions:

   1. Alopecia and neuropathy (must have resolved to ≤ Grade 2)
   2. Congestive Heart Failure (must have been ≤ Grade 1 in severity at the time of occurrence and must have resolved completely)
   3. Anemia (must have resolved to ≤ Grade 2)
8. Patients who have had a last dose of IV chemotherapy within 21 days, last dose of oral cytotoxic chemotherapy, radiotherapy, biological therapy, or investigational therapy within 14 days prior to treatment start. This does not apply to patients already under tucatinib who continue without interruption.
9. Patients who have had any major surgery within 28 days prior to inclusion.
10. Have evidence within 2 years of the start of study treatment of another malignancy that required systemic treatment. This does not apply to patients already under tucatinib who continue without interruption.
11. Concomitant use of other agents for the treatment of cancer or any investigational agent(s).
12. Women who are either pregnant, lactating, planning to get pregnant
13. Have a serious concomitant systemic disorder (eg, active infection or a gastrointestinal disorder causing clinically significant symptoms such as nausea, vomiting, diarrhea, or profound immune suppression) that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol, including but not limited to the following:

    1. Have known human immunodeficiency virus (HIV) infection.
    2. Active hepatitis B or C virus infection (screening required) or have other known chronic liver disease
    3. Severe renal impairment, interstitial lung disease (ILD), severe dyspnea at rest or requiring oxygen therapy, liver disease diagnosed with Child-Pugh A or higher cirrhosis or history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in clinically significant diarrhea.
14. Have clinically significant cardiopulmonary disease such as:

    * ventricular arrhythmia requiring therapy,
    * uncontrolled hypertension (defined as persistent systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications), or
    * any history of symptomatic CHF
    * severe dyspnea at rest (CTCAE Grade 3 or above) due to complications of advanced malignancy
    * hypoxia requiring supplementary oxygen therapy except when oxygen therapy is needed only for obstructive sleep apnea
    * presence of ≥ Grade 2 QTc prolongation on screening ECG
    * conditions potentially resulting in drug-induced prolongation of the QT interval or torsade de pointes:

1. Congenital or acquired long QT syndrome 2. Family history of sudden death 3. History of previous drug induced QT prolongation 4. Current use of medications with known and accepted associated risk of QT prolongation (see row "Accepted Association" in Appendix 8 15. Have known myocardial infarction or unstable angina within 6 months prior to first dose of study treatment 16. Require therapy with warfarin or other coumarin derivatives (non-coumarin anticoagulants are allowed) 17. Have inability to swallow pills or significant gastrointestinal disease which would preclude the adequate oral absorption of medication 18. Patients with altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient informed consent.

19. Person deprived of liberty or placed under a legal protection regime with representation of the person.

20. Inability to comply with medical monitoring of the trial for geographic, social or psychological reasons.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-12-19 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR | 6 months
  The objective response rate (ORR) is defined as the best response defined as complete or partial response occurring within the first 6 months of treatment, assessed by the investigators (according to RECIST v1.1 criteria)

SECONDARY OUTCOMES:
Serious adverse events | From inclusion until 30 days after the last dose of IMP, up to 24 months
  Serious adverse events (SAEs)according to NCI CTCAE v5.0, by grade and their relationship to tucatinib-Oral VP16-trastuzumab.
Adverse events | From inclusion until 30 days after the last dose of IMP, up to 24 months
  Adverse events (AEs) according to NCI CTCAE v5.0, by grade and their relationship to tucatinib-Oral VP16-trastuzumab.
Progression free survival | From inclusion until Progression or Death, up to 24 months
  Progression free survival (PFS) is defined as the time from the date of inclusion until progression per RECIST 1.1 as assessed by the investigator at local site or death due to any cause. The measure of interest is the median PFS
Overall survival | From inclusion until Progression or Death, up to 24 months
  Overall survival (OS) is defined as the time from inclusion to the date of death due to any cause. The measure of interest is the median OS (if reached).
Duration of response | From inclusion until Progression or Death, up to 24 months
  Duration of response (DoR) as defined as the time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by the investigator at local site or death due to any cause. The measure of interest is the median DoR
Time to response | 6 months
  Time to response (TTR) as defined as the time from the start of treatment to the first ORR observed for patients who achieved a CR or PR. The measure of interest is the median TTR.
Clinical benefit rate | 6 months
  Clinical benefit rate (CBR) is defined as the percentage of patients with CR, PR, or stable disease (SD) according to RECIST 1.1, as assessed by the investigator at the local site. The measure of interest is CBR at 24 weeks
EQ-5D-5L scale | From inclusion until Progression or Death, up to 24 months
  The measure of interest is the mean difference in the change from baseline in EQ-5D-5L scale. Time to deterioration in pain, physical functioning, role functioning and global health status/QoL. The EQ VAS score is rated on a scale of 0-100 points. 0 points correspond to the worst possible health status

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément Bidard, Principal Investigator — Institut Curie
Locations (13):
- France (13):
  - Centre Jean Perrin, Clermont-Ferrand, Clermont Ferrand
  - CHU Amiens Picardie-Site Sud, Amiens
  - Institut Sainte Catherine, Avignon
  - Centre François Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut Du Cancer Montpellier, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Institut Curie, Paris
  - Hopital Saint-Louis Ap-Hp Senopole, Paris
  - Centre CARIO-Hôpital Privé des Côtes d'Armor (HPCA), Plérin
  - Institut Curie, Saint-Cloud
  - Oncopole Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).